CLINICAL TRIAL: NCT05844085
Title: Effects of Oat and Oat Components on Cardiometabolic- and Cognitive Test Variables
Brief Title: Effects of Plant-based Polar Lipids on Acute and Second Meal Glucose Tolerance and Appetite Sensations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Anne Nilsson, Associate professor, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Prot.2018/8-Dnr.2018/658
Record Dates: First submitted 2023-04-04; First posted 2023-05-06 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Healthy Subjects; Diet Intervention

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, crossover trial
Who Masked: Participant
Masking Description: the test meals have similar appearance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non-polar lipids (Sham Comparator): A food product containing 15 g plant-based non-polar lipids. The fat is consumed blended with a carbohydrate source containing 50 g available carbohydrates.
  Interventions: Other: Non-polar lipids
- No Lipids (Placebo Comparator): Reference product. A carbohydrate source containing 50 g available carbohydrates.
  Interventions: Other: No lipids
- Polar Lipids low (Experimental): A food product containing 15 g plant-based lipids, of which 50% is polar lipids and 50% is non-polar lipids.The fat is consumed blended with a carbohydrate source containing 50 g available carbohydrates.
  Interventions: Dietary Supplement: Polar lipids low
- Polar Lipids high (Experimental): A food product containing 15 g plant-based lipids, of which 100 % is polar lipids. The fat is consumed blended with a carbohydrate source containing 50 g available carbohydrates.
  Interventions: Dietary Supplement: Polar lipids high

INTERVENTIONS:
Other: Non-polar lipids — The shame comparator lipid intervention product contains no polar lipids. The lipids are mixed with a defined amount of glucose and a flavor enhancer and formulated as a spread. The topping is spread on a defined amount of white wheat bread. The total amounts of lipids are15g, and the total amounts of available carbohydrates are 50 g.
  Arms: Non-polar lipids
Other: No lipids — The placebo comparator contains no added lipids. The product contains a defined amount of glucose and a flavor enhancer and formulated as a spread. The topping is spread on a defined amount of white wheat bread. The total amounts of available carbohydrates are 50 g.
  Arms: No Lipids
Dietary Supplement: Polar lipids low — The experimental intervention product contains 7,5 g plant based lipids polar lipids and 7.5 g plant based lipids non polarlipids. The lipids are mixed with a defined amount of glucose and a flavor enhancer and formulated as a spread. The topping is spread on a defined amount of white wheat bread. TThe total amounts of available carbohydrates are 50 g.
  Arms: Polar Lipids low
Dietary Supplement: Polar lipids high — The experimental intervention product contains15 g plant based polar lipids. The lipids are mixed with a defined amount of glucose and a flavor enhancer and formulated as a spread. The topping is spread on a defined amount of white wheat bread. The total amounts of available carbohydrates are 50 g.
  Arms: Polar Lipids high

SUMMARY:
The overall goal of the project is to increase knowledge which can be used for the development of food products with anti-diabetic properties, with the purpose to facilitate healthier food choices for people. More specifically the primary purpose is to evaluate effects on cardiometabolic test markers of bioactive compounds in healthy humans. Previously the investigators reported beneficial effects of oat polar lipids on cardiometabolic risk markers. In this study the effects previously observed will be compared with cardiometabolic effects of another plant based lipid.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and women
* non-smokers
* between 20-40 years of age
* BMI between 18,5-30 kg/m2
* No known metabolic disorders or food allergies.
* The test subjects should follow a normal diet in accordance with the Nordic Nutrition Recommendations.

Exclusion Criteria:

* Fasting blood glucose ≥6.1 mmol/L
* Use of antibiotics or probiotics in the last three months or during the study period.
* Smoking
* Blood donation during the last two months and during the study.
* Food allergies or food intolerances
* CVD
* Metabolic diseases
* Inflammatory bowel diseases.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Blood glucose concentration (glucose tolerance) | 5.5 hours. Fasting (time =0), 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes, 210 minutes, 225 minutes, 240 minutes, 255 minutes, 270 minutes, 300 minutes, and 330 minutes.
  Test products will be consumed at breakfast. Blood glucose will be determined repeatedly after the breakfast and also following a standardised lunch. The primary outcome measures are incremental areas under the curve after the test breakfast and after the standardised lunch

SECONDARY OUTCOMES:
Subjective hunger sensations | 5.5 hours. Fasting (time =0), 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes, 210 minutes, 225 minutes, 240 minutes, 255 minutes, 270 minutes, 300 minutes, and 330 minutes.
  Test products will be consumed at breakfast. Subjective appetite variables will be determined repeatedly after the breakfast and also following a standardised lunch. The secondary outcome measures are areas under the curve after the test breakfast and after the standardised lunch. Subjective appetite variables will be determined using a 100 mm Visual Analogue Scale (VAS).
Subjective satiety sensations | 5.5 hours. Fasting (time =0), 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes, 210 minutes, 225 minutes, 240 minutes, 255 minutes, 270 minutes, 300 minutes, and 330 minutes.
  Test products will be consumed at breakfast. Subjective appetite variables will be determined repeatedly after the breakfast and also following a standardised lunch. The secondary outcome measures are areas under the curve after the test breakfast and after the standardised lunch. Subjective appetite variables will be determined using a 100 mm Visual Analogue Scale (VAS).
Subjective sensations of desire to eat | 5.5 hours. Fasting (time =0), 15 minutes, 30 minutes, 45 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes, 210 minutes, 225 minutes, 240 minutes, 255 minutes, 270 minutes, 300 minutes, and 330 minutes.
  Test products will be consumed at breakfast. Subjective appetite variables will be determined repeatedly after the breakfast and also following a standardised lunch. The secondary outcome measures are areas under the curve after the test breakfast and after the standardised lunch. Subjective appetite variables will be determined using a 100 mm Visual Analogue Scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- The Human Trial Facility, Food Technology, Engineering and Nutrition, LTH, Lund University, Lund, Välj..., Sweden

IPD SHARING:
Plan to Share IPD: No